CLINICAL TRIAL: NCT01726361
Title: Multidimensional Treatment Foster Care for Adolescents
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: We were not able to recruit families
Sponsor: VIVE - The Danish Center for Social Science Research (Other)
Collaborators: National Board of Social Services, Denmark (Unknown); Ministry of Social Affairs, Denmark (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFI 2506
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Adolescent Behaviour; Family Functioning
Keywords: Multidimension Treatment Foster Care; Adolescents; Disadvantaged families; Out-of-home placement; Conduct Disorder; Family program; Denmark; Youth
MeSH Terms: conditions — Conduct Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MTFC (Experimental): Out of home placement in MTFC family program
  Interventions: Behavioral: Multidimensional Treatment Foster Care
- TAU (Active Comparator): Other kind of out of home placement
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Multidimensional Treatment Foster Care — Out of home placement in MTFC family for 10-12 months
  Arms: MTFC
Behavioral: Treatment as usual — Other kinds of out of home placement
  Other Names: TAU
  Arms: TAU

SUMMARY:
The purpose of the study is to examine the effects of Multidimensional Treatment Foster Care compared to treatment as usual (TAU) for adolescents in Denmark in need of out-of-home placement.

DETAILED DESCRIPTION:
It is difficult to treat adolescents with serious behaviour problems. Although the number of adolescents displaying serious behaviour problems is limited, they are a serious concern to the society e.g. because of their frequent violent behaviour, criminal activities and lack of school adherence.

Multidimensional Treatment Foster Care (MTFC)is a community-based treatment program developed in USA. The goal of the MTFC program is to decrease problem behaviour and to increase developmentally appropriate normative and prosocial behavior in adolescents who are in need of out-of-home placement.

This study will evaluate the effect of MTFC on adolescents in out-of-home placement.

Participants will be recruited by caseworkers in the municipalities and randomly assigned to either MTFC or TAU. TAU will consist of other kinds of out-of-home placements. Outcomes will be assessed for all participants at baseline, post-treatment (12 months), and 12 months post-treatment. Parents and youth will be asked to fill out questionnaires on e.g. behaviour, parental stress, sense of cohesion, general health.

ELIGIBILITY:
Inclusion Criteria:

* 12-17 years old
* In need of out of home placement
* serious behaviour problems

Exclusion Criteria:

* severe psychiatric illness in youth or parent
* risk of suicide in youth
* acute psychosis in youth
* sexual offence by youth
* severe substance abuse in youth or parent

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Strengths and difficulties questionnaire, Child Behavior Checklist | 12 months post baseline
  Measuring child/youth behaviour

SECONDARY OUTCOMES:
Parental Stress Scale | 12 months post baseline
  Measuring parental stress
Sense of Cohesion 13 | 12 months post baseline
  Measuring stress in human functioning
Ladder of life | 12 months post baseline
  Measuring overall quality of life
Major Depression Index 10 | 12 months post baseline
  Measuring parent's depression symptoms

OTHER OUTCOMES:
Other outcomes | 12 months post baseline
  crime (register and self-report) school truancy (register and self-report) general health including substance abuse (self-report)

CONTACTS AND LOCATIONS:
Overall Officials: Mette Deding, Study Director — SFI the Danish National Centre for Social Research
Locations (1):
- SFI the Danish National Centre for Social Research, Copenhagen, Denmark